CLINICAL TRIAL: NCT01837134
Title: TeleLifestyleCoaching Study - Telemedical Coaching for Weight Loss
Brief Title: Telemedical Coaching for Weight Loss
Acronym: Fit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West German Center of Diabetes and Health (Other)
Responsible Party: Principal Investigator, Stephan Martin, Director of the West German Center of Diabetes and Health, West German Center of Diabetes and Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Telemedical coaching; 98149 (Other Grant/Funding Number: Boehringer Ingelheim Pharma GmbH & Co.KG)
Record Dates: First submitted 2013-04-15; First posted 2013-04-22 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Overweight; Obesity; Metabolic Syndrome
Keywords: telemedicine; overweight; obesity
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome | interventions — Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (C) group (No Intervention): The control group will remain in routine care for 12 weeks. After 12 weeks they will also be given a weighing machine and a step counter, with automatic transfer into a personalized online portal, which can be monitored from both, the participant and the study centre. During the next 12 weeks they will get care calls from the study centre aiming to discuss measured data and to fix target agreements.
- telemedical (TM) group (Experimental): Participants in the telemedical (TM) group will get a weighing machine and a step counter, with automatic transfer into a personalized online portal, which can be monitored from both, the participant and the study centre.
  Interventions: Device: telemedical (TM) group
- telemedical coaching (TMC) group (Experimental): Participants in the telemedical coaching (TMC) group will get a weighing machine and a step counter, with automatic transfer into a personalized online portal, which can be monitored from both, the participant and the study centre. Additionally, they will be called once per week for 12 weeks from the study centre aiming to discuss measured data and to fix target agreements. After 12 weeks the care calls be be given once per month for further 9 months.
  Interventions: Device: telemedical (TM) group; Behavioral: telemedical coaching (TMC) group

INTERVENTIONS:
Device: telemedical (TM) group — telemedical devices (weighing machine and step counter)
  Arms: telemedical (TM) group; telemedical coaching (TMC) group
Behavioral: telemedical coaching (TMC) group — care calls once per week for 12 weeks
  Arms: telemedical coaching (TMC) group

SUMMARY:
Lifestyle changes often fail due to loss of motivation. Telemedicine and personal coaching have the potential to support lifestyle change and weight loss. Therefore, the aim of our randomized controlled trial is to examine the effect of telemedicine with and without coaching in comparison to a control group on weight loss in overweight participants.

DETAILED DESCRIPTION:
In an occupational health care setting employees with overweight and/or metabolic syndrome will be randomized into a three arm 12-week trial. Participants in the telemedical (TM) and telemedical coaching (TMC) group got a weighing machine and a step counter, with automatic transfer into a personalized online portal, which could be monitored from both, the participant and the study centre. The TMC group weekly will get care calls from the study centre aiming to discuss measured data and to fix target agreements. The control group will remain in routine care.

ELIGIBILITY:
Inclusion Criteria:

* employed at Boehringer Ingelheim Pharma GmbH for at least 2 years
* older than 40 years
* overweight or obese or metabolic syndrome

Exclusion Criteria:

* not willing to participate

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
weight loss | 12 weeks
  Weight will be measured at baseline and after 12 weeks.

SECONDARY OUTCOMES:
cardiometabolic risk factors | 12 weeks
quality of life | 12 weeks
  Quality of life will be assessed by the validated questionnaires ADS-L and SF-12.
physical activity | 12 weeks
  Physical activity will be assessed using a validated questionnaire.

OTHER OUTCOMES:
eating behaviour | 12 weeks
  Eating behaviour will be measured using the validated questionnaire FEV.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Martin, MD, Principal Investigator — West-German Centre of Diabetes and Health
Locations (1):
- West-German Centre of Diabetes and Health, Düsseldorf, Germany

REFERENCES:
- [Derived] Kempf K, Rohling M, Martin S, Schneider M. Telemedical coaching for weight loss in overweight employees: a three-armed randomised controlled trial. BMJ Open. 2019 Apr 11;9(4):e022242. doi: 10.1136/bmjopen-2018-022242. PMID 30975666